CLINICAL TRIAL: NCT01160471
Title: Noninvasive Imaging of Heart Failure
Brief Title: Noninvasive Imaging of Heart Failure: A Pilot Study
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 100153; 10-CC-0153
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-10-30

CONDITIONS: MRI; Acquired Heart Disease; Myocardial Fibrosis
Keywords: Heart Failure; MRI; Ultrasound; Fibrosis; Biomarker
MeSH Terms: conditions — Heart Failure; Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Healthy Volunteers: Adult men and women without a clinical diagnosis of heart failure
- Patients: Adult men and women with a clinical diagnosis of heart failure

SUMMARY:
Background:

- Heart failure is a common cardiovascular disorder whose incidence increases with age, affecting up to 10% of people older than 65 years of age. As the population ages, the prevalence and cost of heart failure will continue to rise. Researchers are interested in using noninvasive imaging methods to better understand the symptoms and effects of heart failure.

Objectives:

- To conduct a noninvasive comparative imaging study of individuals with heart failure.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with heart failure (with at least mild symptoms and slight limitations on physical activity).

Design:

* This study will last approximately 2 years and will require four visits to the National Institutes of Health Clinical Center, with one screening visit and three study visits.
* Participants will be screened with a full medical history and physical examination, as well as blood and urine samples.
* Participants will have the following tests during each study visit:
* Physical examination
* Blood and urine samples
* Cardiac magnetic resonance imaging
* Cardiac computerized tomography to study the blood vessels in and leading to the heart
* Echocardiogram to evaluate heart function
* Electrocardiogram to measure heart electrical activity
* The three study visits will take place 1 year apart. Participants will also receive follow-up phone calls 6 months after the first and second visits.
* No treatment will be provided as part of this protocol.

DETAILED DESCRIPTION:
More than 9% of American men and close to 5% of women ages 60 to 79 years report a diagnosis of heart failure, where above the age of 80 years these figures increase to 13.8% and 12.2%, respectively. Projection into the middle part of this century suggests that, as the population ages, the prevalence and cost of heart failure will continue to rise. The primary aim of this proposal is to investigate noninvasive imaging methods for quantifying diffuse myocardial fibrosis with cardiac magnetic resonance imaging (CMR) in heart failure patients. The secondary aims are to investigate the association between diffuse fibrosis detected by CMR with left ventricular function, and examine the utility of multi-detector CT (MDCT) in detecting diffusion myocardial fibrosis.

ELIGIBILITY:
* INCLUSION CRITERIA:

The common inclusion criteria between patients and controls are:

A. Able to understand and sign informed consent.

B. Able to complete a MRI or CT scan.

C. Age greater than or equal to 18 years old.

Heart Failure subject:

D. Men and women with a clinical diagnosis of heart failure.

E. New York Heart Association functional class II or worse.

F. For the normal ejection fraction arm.

1. Preserved left ventricular ejection fraction (EF >50%)
2. Diastolic dysfunction defined one or more of the following

   1. LVEDP > 16 mm Hg
   2. PCW > 12 mm Hg
   3. E/E ratio >15
   4. E/E ratio >8 AND NT-proBNP >220 pg/mL

   For the systolic dysfunction arm:
3. Left ventricular ejection fraction <40%

   Normal Control:

   G. Men and women without a clinical diagnosis of heart failure.

   H. NIH employees may be involved and NIH requirements will be followed as laid out in NIH Policy Manual 2300-630-3 - Leave Policy For NIH Employees Participating In NIH Medical Research Studies.

   EXCLUSION CRITERIA:

   Individuals will be excluded from the study if they are discovered to have coexistent conditions that may contribute to structural or functional cardiac abnormalities, which may confound interpretation of results, are ineligible for MRI or if they are at increased risk for Nephrogenic Systemic Fibrosis (NSF) including:

   A. Contra indications for gadiolinium-based contrast agent:
   1. eGFR < 30ml/min/1.73m(2)
   2. Acute renal failure, renal transplantation, current dialysis treatment or hepatorenal syndrome
   3. History of liver transplantation or severe liver disease
   4. Severe Asthma
   5. Hemoglobinopathies, sickle cell anemia and thalassemias major
   6. History of multiple myeloma
   7. History of significant allergic reaction to gadolinium-based contrast agents

   B. Medical conditions associated with increased collagen turnover which may confound interpretation of biomarkers of collagen synthesis. Examples include systemic amyloid disease, cirrhosis, liver, pulmonary, or renal fibrosis, inflammatory states, cancer, recent trauma or surgery;

   C. Pregnant or lactating women;

   D. Mental, neurologic or social condition preventing understanding of the rationale, procedures, risks and potential benefits associated with the trial;

   E. Any other conditions that precludes safety for MRI or MDCT per the researcher s evaluation.

   F. Patients otherwise eligible but with any of the following contraindications for iodine-based CT contrast agent will be excluded from contrast CT angiography but may undergo all other study procedures:
   1. Renal dysfunction (defined as eGFR <45 mL/min/m(2))
   2. Current clinical diagnosis of renal failure
   3. Prior hypersensitivity to iodine containing substances (shellfish, iodine, and or previous contrast reactions to contrast agents.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2010-07-01; Study Completion 2019-10-30

PRIMARY OUTCOMES:
Post contrast myocardial T1 measured by CMR. | Study end
  The primary aim of this protocol is to investigate noninvasive imaging methods for quantifying diffuse myocardial fibrosis with cardiac magnetic resonance imaging(CMR) in heart failure patient

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Jones, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Nacif MS, Liu Y, Yao J, Liu S, Sibley CT, Summers RM, Bluemke DA. 3D left ventricular extracellular volume fraction by low-radiation dose cardiac CT: assessment of interstitial myocardial fibrosis. J Cardiovasc Comput Tomogr. 2013 Jan-Feb;7(1):51-7. doi: 10.1016/j.jcct.2012.10.010. Epub 2012 Dec 4. PMID 23333188